CLINICAL TRIAL: NCT05064930
Title: Assessment of the Efficacy of Single-strain Probiotics in Patients With Irritable Bowel Syndrome - a Randomized Double-blind Placebo-controlled Study
Brief Title: The Efficacy of Single-strain Probiotics in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordic Biotic Sp. z o.o. (Industry)
Collaborators: Medical University of Lublin (Other)
Responsible Party: Principal Investigator, Barbara Skrzydło-Radomańska, Profesor, MD, PhD, Nordic Biotic Sp. z o.o.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT/NB/120/2020/PR-SS
Record Dates: First submitted 2021-09-10; First posted 2021-10-01 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Irritable Bowel Syndrome
Keywords: Probiotics
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Bifidobacterium lactis (Active Comparator): Probiotic formula contains 5x109 Bifidobacterium lactis Nordbiotic™ BI040 colony forming units (CFU)/capsule
  Interventions: Dietary Supplement: Probiotic Bifidobacterium lactis
- Bacillus coagulans (Active Comparator): Probiotic formula contains 2x109 Bacillus coagulans Nordbiotic™BC300 colony forming units (CFU)/capsule
  Interventions: Dietary Supplement: Probiotic Bacillus coagulans
- Maltodextrin (Placebo Comparator): Maltodextrin (starch hydrolisate) as a compound presents in probiotic formula.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic Bifidobacterium lactis — The probiotic will be administered orally over a period of 12 weeks.
  Arms: Bifidobacterium lactis
Dietary Supplement: Probiotic Bacillus coagulans — The probiotic will be administered orally over a period of 12 weeks.
  Arms: Bacillus coagulans
Dietary Supplement: Placebo — Maltodextrin as a placebo will be administered orally over a period of 12 weeks. The taste and appearance of the placebo will be similar to those of the probiotic formulation.
  Arms: Maltodextrin

SUMMARY:
Irritable bowel syndrome (IBS) is one of the most common, yet still not fully understood, gastrointestinal disorders in adults. One suspected etiology involves intestinal dysbiosis, i.e. both quantitative and qualitative alterations in intestinal microbiota composition, which affects the gut-brain axis. Probiotics are live microorganisms, which-administered at the right dose-are beneficial for human health; their mechanism of action involves modifying the gut microbiota. Clinical study reports document that probiotic administration is beneficial for patients with IBS. The ultimate clinical effects depend primarily on probiotic strain selection. Our research team evaluated a multi-strain probiotic formulation and a multi-strain synbiotic (a combination of probiotic strains with short-chain prebiotic fructooligosaccharides) formulation as part of two randomized placebo-controlled clinical trials in patients with IBS with predominant diarrhea. The results indicated a beneficial effect of these formulations on the clinical course of IBS assessed with the international IBS symptom severity scale (IBS-SSS), with each of the study formulations exhibiting efficacy in different fields. The formulation composed of a mixture of Bifidobacterium and Lactobacillus strains reduced the levels of pain and improved the quality of life, whereas the synbiotic formulation effectively improved bloating and had a beneficial effect on the general condition of the intestines. A systematic review and meta-analysis published in 2020 showed that high doses of single-strain formulations, particularly those containing Bifidobacterium or Lactobacillus strains, may be more effective in IBS patients. Other reports demonstrated a high efficacy of the new-generation probiotic Bacillus coagulans in IBS. Therefore, the main objective of this research project is to assess the efficacy of single-strain probiotics containing Bifidobacterium lactis or Bacillus coagulans in patients with IBS.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo-controlled trial included 120 adult patients, who had been diagnosed with IBS according to the Rome IV diagnostic criteria. The patients will receive orally a probiotic formulation containing Bifidobacterium lactis or Bacillus coagulans or placebo over a period of 12 weeks. Once the period of supplementation is completed, the patients will be followed-up for the subsequent 4 weeks. The patients included in the study will receive diaries, which they will complete daily. The patient's dairy will include information about the number of stools, stool consistency (assessed based on the Bristol Stool Form Scale) and IBS symptoms (abdominal pain, bloating, bowel urgency, and feeling of incomplete evacuation) rated in a 5-grade scale. The diary will also include information on any adverse events and the use of any new medications during the study. Once a week, the patients will be contacted by phone by interviewers who will collect the information recorded in the patient's diary.

During the first visit, the patients included in the study will be informed of the study procedure and educated on the phone exchanges with the interviewers. One week prior to study intervention, the patients will be asked to record their symptoms in their patient diaries every day. Subsequently, the patients will visit their study doctor every four weeks (from the beginning of the study intervention) in order to receive the next dose of the study formulation/placebo. During each study visit, the patients will be evaluated with the use of IBS-SSS and IBS Global Improvement Scale (IBS-GIS). The patients included in the study will undergo a hydrogen breath test for small intestinal bacterial overgrowth (SIBO) both prior to receiving the study formulation/placebo and 12 weeks later, after intervention is completed.

The study will last a total of 16 weeks from the moment the intervention is initiated (12 weeks of interventions and 4 weeks of follow-up).

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian males and females;
2. Age from 18 to 70 years, inclusive;
3. Good physical and mental condition assessed based on the patient's history and physical examination;
4. Laboratory test results (blood tests, including blood chemistry and antibody tests; and urinalysis) within the normal limits for the local laboratory or considered clinically insignificant by the study investigator;
5. A voluntarily provided written informed consent;
6. Being available throughout the duration of the study;
7. Patients with IBS diagnosed based on the Rome IV criteria;
8. Patients with any form of IBS of at least moderate severity assessed via the IBS-SSS (score >175).

Exclusion Criteria:

1. Cardiovascular disorders: uncontrolled hypertension (blood pressure > 170/100 mmHg), cerebrovascular disease;
2. Severe respiratory disorders (asthma, chronic obstructive pulmonary disease)
3. Liver or kidney disease and unexplained blood chemistry abnormalities: serum creatinine of more than twice the upper limit of normal, serum aminotransferease (AST or ALT) levels more than twice the upper limit of normal;
4. Gastrointestinal disorders other than IBS (including gastroenteritis, celiac disease, and bacterial infections or parasitic infestations confirmed either clinically or endoscopically);
5. Endocrine disorders, including diabetes (fasting blood glucose > 11 mmol/L) and serum thyroid stimulating hormone (TSH) levels above normal;
6. Severe neurological conditions, with psychosis;
7. Malignancy;
8. Pregnancy or breastfeeding;
9. Hypersensitivity to soy;
10. Lactose intolerance that may explain the symptoms (i.e. the symptoms resolve or considerably subside in response to a lactose-free diet);
11. The use of gastrointestinal motility stimulants or dietary fiber supplements during the 2 weeks preceding the clinical study;
12. The use of antithrombotic agents;
13. A surgical procedure scheduled during the course of the clinical study;
14. Current probiotic use and refusal to undergo a 3-month washout period;
15. Antibiotic therapy within the previous 3 months;
16. The patients who receive antibiotics during the study will be excluded;
17. Being included in another clinical study within the previous 3 months;
18. History of alcohol or substance abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in severity of IBS symptoms using IBS Severity Scoring System (IBS-SSS) | From baseline at 4, 8, 12 weeks of intervention, and 4 weeks (16 weeks of the study) after intervention
  IBS-SSS is a 5-question survey that asks: 1. the severity of abdominal pain, 2. frequency of abdominal pain, 3. severity of abdominal distention, 4.dissatisfaction with bowel habit, and 5. interference with quality of life over the past 10 days. Subjects respond to each question on a 100-point visual analogue scale. Each of the five question generates a maximum score of 100 point, and total scores can range from 0-500 with higher scores indicating severe symptoms. A decrease of 50 points is associated with a clinically meaningful improvement.
Improvement of IBS global symptoms using Global Improvement Scale (IBS-GIS) | From baseline at 4, 8, 12 weeks of intervention, and 4 weeks (16 weeks of the study) after intervention
  IBS-Global Improvement Scale assesses IBS symptoms using a patient-defined 7 point Likert scale ranging from symptoms substantially worse to substantially improved.
  Patients answer the question "Have you felt any change in the severity of your symptoms over the past 7 days compared to how you felt before the medicine was given?
  The answers are recorded based on the 7-point scale:
  1. = I feel that the symptoms have worsened significantly
  2. = I feel that the symptoms have moderately worsened
  3. = I feel that the symptoms have slightly worsened
  4. = I feel no change
  5. = I feel a slight improvement
  6. = I feel moderate improvement
  7. = I feel significant improvement IBS-GIS score indicates: improvement if is >4 or worsening if is<4, no change if is 4

SECONDARY OUTCOMES:
Changes in number of stools | From baseline for 12 weeks of intervention, and for 4 weeks after intervention
  The number of stools per day assessed before intervention and then 3 times a week
Changes in severity of pain | From baseline for 12 weeks of intervention, and for 4 weeks after intervention
  The severity of pain assessed before intervention and then 3 times a week using a patient-defined 5 point Likert scale: point 0 - no pain, and 1-4 the severity of pain with higher scores indicating worse pain.
Changes in flatulence | From baseline for 12 weeks of intervention, and for 4 weeks after intervention
  The severity of flatulence assessed before intervention and then 3 times a week using a patient-defined 5 point Likert scale: point 0 - no flatulence/abdominal distension, and 1-4 the severity of flatulence/abdominal distension with higher scores indicating worse pain.
Occurrence of side effects | From baseline for 12 weeks of intervention
  Side effects will be pointed in patient's dairy and collected by phone by interviewers.
Changes in type of stools | From baseline for 12 weeks of intervention, and for 4 weeks after intervention
  The type of stools analyzed before intervention and then 3 times a week. Type of stools assessed using the Bristol Stool Scale (BSS). BSS is designed to classify faeces into seven groups: type 1-2 indicate constipation, type 3-4 are "normal" stools; type 5-7 indicate diarrhea. The type of stool will be assessed with 7-point numerical scale (range 1-7).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Skrzydło-Radomańska, MD, PhD, Principal Investigator — Medical University of Lublin
Locations (1):
- Medical University of Lublin, Lublin, Poland

REFERENCES:
- [Derived] Skrzydlo-Radomanska B, Prozorow-Krol B, Kurzeja-Miroslaw A, Cichoz-Lach H, Laskowska K, Majsiak E, Bierla JB, Agnieszka S, Cukrowska B. The Efficacy and Safety of Single-Strain Probiotic Formulations Containing Bifidobacterium lactis or Bacillus coagulans in Adult Patients with Irritable Bowel Syndrome-A Randomized Double-Blind Placebo-Controlled Three-Arm Interventional Trial. J Clin Med. 2023 Jul 22;12(14):4838. doi: 10.3390/jcm12144838. PMID 37510953